CLINICAL TRIAL: NCT01377220
Title: Evaluation of 11 C-Choline PET-CT for Detection of Hepatocellular Carcinoma
Acronym: CHOLPET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Commissariat A L'energie Atomique (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: CASTILLA-LIEVRE Maria-Angéla, MD, Assistance Publique - Hôpitaux de Paris
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-020221
Record Dates: First submitted 2011-06-07; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Positron Emission Tomography/computed tomography (PET-CT); 11C-Choline; alpha fetoprotein; Dynamic magnetic resonance imaging; Abdomen computed tomography; Tumoral liver biopsy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 11C-Choline — 11C-Choline : 6MBq/kg on direct intravenous on one minute.

SUMMARY:
Hepatocellular carcinoma (HCC)is the most frequent primitive tumour of the liver.

Recently, several research studies reported that 11C-choline PET has shown a high detection rate of well differentiated HCC, which is an early stage of primary liver cancer. The aim of this study was to prospectively evaluate the diagnostic accuracy of 11C-choline PET-CT to detect HCC in cirrhotic or non cirrhotic patients.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC)is the most frequent primitive tumour of the liver. Although the histological examination remains the reference for the diagnosis, it may be difficult to obtain biopsy material because of difficulty in getting to the lesion or due to their small size. However, it is know that the size of the lesion remains a major prognostic factor, implying the need for an earliest detection, which enhances the chance for curative treatment.PET enables the study of changes in the glucidic or lipidic metabolism of cancer cells. PET-CT, providing both metabolic and anatomic information, improves the performances of this technique. PET with 18F-FDG has not been sensitive enough in the detection of HCC, except in cases of low grade. Recently, several research studies reported that 11C-choline PET has shown a high detection rate of well differentiated HCC, which is an early stage of primary liver cancer.

The study include 30 patients presenting a suspicion of HCC with or without cirrhosis. Each patient will be examined with two conventional imaging techniques, consisting in dynamic magnetic resonance imaging and computed tomography; alpha fetoprotein measurement will be taken. PET-CT will be acquired after an intravenous injection of 11C-choline. The 11C-choline PET-CT performance for HCC diagnosis will be compare to histological analysis obtained by a tumoral liver biopsy, or by using of the American Association for the study of Liver Disease diagnostic criteria. In absence of the two criteria , the follow up within one year will serve as a reference.

ELIGIBILITY:
Inclusion Criteria:

* Patients up to 18 years old with
* Patients with suspicion hepatocellular carcinoma on conventional imaging(hepatic ultrasonography, abdominal computed tomography, dynamic resonance magnetic)and/or on alpha fetoprotein measurement
* Patients with suspicion recurrence of hepatocellular carcinoma on conventional imaging(hepatic ultrasonography, abdominal computed tomography, dynamic resonance magnetic)and/or on alpha fetoprotein measurement
* Patients which perform two conventional imaging techniques, consisting in dynamic magnetic resonance imaging (MRI) and computed tomography (CT)and must have an alpha fetoprotein measurement
* Patients which perform 18F-FDG PET-CT
* Informed Consent Form signed and dated by patients
* Patients which are "Security Social" affiliated

Exclusion Criteria:

* Pregnant or suckling women
* Women able to procreate, without efficient birth control
* Patients with an other tumoral disease
* Patients with chemotherapy or surgery from less than four weeks
* Patients with radiotherapy from less four months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Angéla M-A CASTILLA-LIEVRE, MD, Principal Investigator — Hôpital Antoine Béclère 92140 CLAMART-FRANCE
Locations (1):
- CEA-SHFJ, Orsay, France

REFERENCES:
- [Background] Talbot JN, Fartoux L, Balogova S, Nataf V, Kerrou K, Gutman F, Huchet V, Ancel D, Grange JD, Rosmorduc O. Detection of hepatocellular carcinoma with PET/CT: a prospective comparison of 18F-fluorocholine and 18F-FDG in patients with cirrhosis or chronic liver disease. J Nucl Med. 2010 Nov;51(11):1699-706. doi: 10.2967/jnumed.110.075507. Epub 2010 Oct 18. PMID 20956466
- [Background] Tolvanen T, Yli-Kerttula T, Ujula T, Autio A, Lehikoinen P, Minn H, Roivainen A. Biodistribution and radiation dosimetry of [(11)C]choline: a comparison between rat and human data. Eur J Nucl Med Mol Imaging. 2010 May;37(5):874-83. doi: 10.1007/s00259-009-1346-z. Epub 2010 Jan 13. PMID 20069295
- [Background] Park JW, Kim JH, Kim SK, Kang KW, Park KW, Choi JI, Lee WJ, Kim CM, Nam BH. A prospective evaluation of 18F-FDG and 11C-acetate PET/CT for detection of primary and metastatic hepatocellular carcinoma. J Nucl Med. 2008 Dec;49(12):1912-21. doi: 10.2967/jnumed.108.055087. Epub 2008 Nov 7. PMID 18997056
- [Background] Ho CL, Yu SC, Yeung DW. 11C-acetate PET imaging in hepatocellular carcinoma and other liver masses. J Nucl Med. 2003 Feb;44(2):213-21. PMID 12571212
- [Background] Hwang KH, Choi DJ, Lee SY, Lee MK, Choe W. Evaluation of patients with hepatocellular carcinomas using [(11)C]acetate and [(18)F]FDG PET/CT: A preliminary study. Appl Radiat Isot. 2009 Jul-Aug;67(7-8):1195-8. doi: 10.1016/j.apradiso.2009.02.011. Epub 2009 Feb 20. PMID 19342249
- [Background] Talbot JN, Gutman F, Fartoux L, Grange JD, Ganne N, Kerrou K, Grahek D, Montravers F, Poupon R, Rosmorduc O. PET/CT in patients with hepatocellular carcinoma using [(18)F]fluorocholine: preliminary comparison with [(18)F]FDG PET/CT. Eur J Nucl Med Mol Imaging. 2006 Nov;33(11):1285-9. doi: 10.1007/s00259-006-0164-9. Epub 2006 Jun 27. PMID 16802155
- [Background] Yamamoto Y, Nishiyama Y, Kameyama R, Okano K, Kashiwagi H, Deguchi A, Kaji M, Ohkawa M. Detection of hepatocellular carcinoma using 11C-choline PET: comparison with 18F-FDG PET. J Nucl Med. 2008 Aug;49(8):1245-8. doi: 10.2967/jnumed.108.052639. Epub 2008 Jul 16. PMID 18632827
- [Background] Salem N, Kuang Y, Wang F, Maclennan GT, Lee Z. PET imaging of hepatocellular carcinoma with 2-deoxy-2[18F]fluoro-D-glucose, 6-deoxy-6[18F] fluoro-D-glucose, [1-11C]-acetate and [N-methyl-11C]-choline. Q J Nucl Med Mol Imaging. 2009 Apr;53(2):144-56. Epub 2008 Nov 28. PMID 19039303
- [Background] Hara T, Kosaka N, Shinoura N, Kondo T. PET imaging of brain tumor with [methyl-11C]choline. J Nucl Med. 1997 Jun;38(6):842-7. PMID 9189127
- [Background] Hara T, Kosaka N, Kishi H. PET imaging of prostate cancer using carbon-11-choline. J Nucl Med. 1998 Jun;39(6):990-5. PMID 9627331
- [Background] Li CW, Kuo YC, Chen CY, Kuo YT, Chiu YY, She FO, Liu GC. Quantification of choline compounds in human hepatic tumors by proton MR spectroscopy at 3 T. Magn Reson Med. 2005 Apr;53(4):770-6. doi: 10.1002/mrm.20412. PMID 15799049
- [Background] Kojiro M, Roskams T. Early hepatocellular carcinoma and dysplastic nodules. Semin Liver Dis. 2005;25(2):133-42. doi: 10.1055/s-2005-871193. PMID 15918142
- [Background] Kim HO, Kim JS, Shin YM, Ryu JS, Lee YS, Lee SG. Evaluation of metabolic characteristics and viability of lipiodolized hepatocellular carcinomas using 18F-FDG PET/CT. J Nucl Med. 2010 Dec;51(12):1849-56. doi: 10.2967/jnumed.110.079244. PMID 21098794
- [Background] Kim YK, Lee KW, Cho SY, Han SS, Kim SH, Kim SK, Park SJ. Usefulness 18F-FDG positron emission tomography/computed tomography for detecting recurrence of hepatocellular carcinoma in posttransplant patients. Liver Transpl. 2010 Jun;16(6):767-72. doi: 10.1002/lt.22069. PMID 20517911
- [Background] Wolfort RM, Papillion PW, Turnage RH, Lillien DL, Ramaswamy MR, Zibari GB. Role of FDG-PET in the evaluation and staging of hepatocellular carcinoma with comparison of tumor size, AFP level, and histologic grade. Int Surg. 2010 Jan-Mar;95(1):67-75. PMID 20480845
- [Background] Khan MA, Combs CS, Brunt EM, Lowe VJ, Wolverson MK, Solomon H, Collins BT, Di Bisceglie AM. Positron emission tomography scanning in the evaluation of hepatocellular carcinoma. J Hepatol. 2000 May;32(5):792-7. doi: 10.1016/s0168-8278(00)80248-2. PMID 10845666
- [Background] Delbeke D, Martin WH, Sandler MP, Chapman WC, Wright JK Jr, Pinson CW. Evaluation of benign vs malignant hepatic lesions with positron emission tomography. Arch Surg. 1998 May;133(5):510-5; discussion 515-6. doi: 10.1001/archsurg.133.5.510. PMID 9605913
- [Background] Okazumi S, Isono K, Enomoto K, Kikuchi T, Ozaki M, Yamamoto H, Hayashi H, Asano T, Ryu M. Evaluation of liver tumors using fluorine-18-fluorodeoxyglucose PET: characterization of tumor and assessment of effect of treatment. J Nucl Med. 1992 Mar;33(3):333-9. PMID 1311035
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] Bruix J, Sherman M, Llovet JM, Beaugrand M, Lencioni R, Burroughs AK, Christensen E, Pagliaro L, Colombo M, Rodes J; EASL Panel of Experts on HCC. Clinical management of hepatocellular carcinoma. Conclusions of the Barcelona-2000 EASL conference. European Association for the Study of the Liver. J Hepatol. 2001 Sep;35(3):421-30. doi: 10.1016/s0168-8278(01)00130-1. No abstract available. PMID 11592607